CLINICAL TRIAL: NCT01689818
Title: Long-term Follow-up of Functional Performance and Exercise Efficacy in Community-dwelling Elderly With Insomnia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 201012130RB
Record Dates: First submitted 2012-08-28; First posted 2012-09-21 (Estimated); Last update posted 2012-09-21 (Estimated); Status verified 2012-09

CONDITIONS: Insomnia
Keywords: insomnia, elderly, exercise training
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- exercise training (Experimental): exercise training program which included aerobic exercise for 3 times per week.
  Interventions: Other: exercise training
- control (No Intervention): lifestyle counseling

INTERVENTIONS:
Other: exercise training — exercise training program which included aerobic exercise for 3 times per week.
  Arms: exercise training

SUMMARY:
Poor sleep quality has been recognized as a major public health concern in the world. The prevalence of insomnia in Taiwan is comparable to that of Western countries. It is estimated that up to 50% of elderly complain about their sleep. Insomnia is associated with anxiety, falls, or cognitive impairment in the elderly, which may compromise their daily activities function and quality of life.

Recently, researches have demonstrated the associations between insomnia and endocrine system dysfunction, metabolic disorders, and cardiovascular events and death. Therefore, it is an important issue to improve sleep quality of the elders. The side-effects of pharmacological treatments and high-cost of cognitive behavior therapy limit their accessibility and effectiveness, and exercise training has been expected to provide an alternative intervention for insomnia. However, the long-term impact of insomnia on health-related fitness and metabolic function, and the effect of exercise training remain inconclusive. Therefore, the study hypothesis is that exercise training affect functional performance and quality of life in community-dwelling elderly with insomnia.

DETAILED DESCRIPTION:
This project will be conducted in three years:

In the first year, we will compare the cardiorespiratory function, body composition, physical activity, and metabolic biochemistry parameters in community-dwelling elders with good and poor sleep quality. One hundred and twenty elders will be recruited to receive the actigraph accelermometer recording, sleep quality questionnaire, exercise test, bioelectrical impedance analysis, heart rate variability analysis, cognitive and depression evaluation, and biochemistry analysis.

Secondly, the study will evaluate the efficacy and possible mechanisms of a 16-week exercise training for insomnia. Sixty patients with insomnia elders will be randomized to exercise group or control group. Participants in the exercise group will receive aerobic and resistance exercise 3 times per week for 16 weeks. The controls will receive sleep hygiene education and consultation. All measurements will be performed as described before.

Finally, all the 120 elders participating in this study will receive 12-month follow-up assessments to explore the longitudinal impact of insomnia on cardiorespiratory function, body composition and metabolic function, and long-term effect of exercise training on insomnia. We expect elders with poor sleep quality have lower level of health-related fitness and metabolic function; exercise training is effective to improve sleep quality, metabolic function and general health in the elders with insomnia, and the effect can be sustained for a long period.

ELIGIBILITY:
Inclusion Criteria:

* above 65 y/o elderly

Exclusion Criteria:

* psychiatric diagnosis (DSM-IV) of serious mental illness, including severe depression symptoms, mania, Alcohol or drug abuse
* with other sleep disorders such as sleep apnea, periodic limb twitching, or fast moving eye movement behavior disorder
* cognitive and other neurological diseases history who can not communicate
* Unstable serious illness or sports contraindicated cardiopulmonary disease such as diabetes, hypertension, and other cardiovascular disease, neurological injury patients
* body mass index greater than 35 kg/ M 2 or more

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2011-08; Primary Completion 2014-07 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
functional performance | 16 weeks
  physical fitness and physical disability

SECONDARY OUTCOMES:
depression | 16 weeks

OTHER OUTCOMES:
cognitive function | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Meng-Yueh Chien, PhD, Principal Investigator — National Taiwan University
Locations (1):
- Meng-Yueh Chien, Taipei, Taiwan

REFERENCES:
- [Derived] Chien MY, Chen HC. Poor sleep quality is independently associated with physical disability in older adults. J Clin Sleep Med. 2015 Mar 15;11(3):225-32. doi: 10.5664/jcsm.4532. PMID 25515275